CLINICAL TRIAL: NCT06161532
Title: A Phase II Study of Sacituzumab Govitecan With or Without Atezolizumab Immunotherapy in Rare Genitourinary Tumors (SMART) Such as High Grade Neuroendocrine Carcinomas, Adenocarcinoma, and Squamous Cell Bladder/Urinary Tract Cancer, Renal Medullary Carcinoma and Penile Cancer
Brief Title: Sacituzumab Govitecan With or Without Atezolizumab Immunotherapy in Rare Genitourinary Tumors (SMART) Such as High Grade Neuroendocrine Carcinomas, Adenocarcinoma, and Squamous Cell Bladder/Urinary Tract Cancer, Renal Medullary Carcinoma and Penile C...
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001535; 001535-C
Record Dates: First submitted 2023-12-02; First posted 2023-12-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11-24

CONDITIONS: Small Cell Carcinoma of the Bladder; Small Cell Carcinoma of the Urinary Tract; Squamous Cell Carcinoma of the Bladder; Squamous Cell Carcinoma of the Urinary Tract; Primary Adenocarcinoma of the Bladder; Primary Adenocarcinoma of the Urinary Tract; Renal Medullary Carcinoma; Squamous Cell Carcinoma of the Penis
Keywords: Urothelial carcinoma; Trophoblastic cell surface antigen 2; Programmed death-ligand 1; SN-38; Immunotherapy
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — sacituzumab govitecan; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Treatment with sacituzumab govitecan
  Interventions: Drug: Sacituzumab govitecan
- Arm 2 (Experimental): Treatment with sacituzumab govitecan and atezolizumab
  Interventions: Drug: Sacituzumab govitecan; Drug: Atezolizumab

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab govitecan is administered IV at 10 mg/kg on days 1 and 8 of each 21-day cycle.
Drug: Atezolizumab — Atezolizumab is administered IV at 1200 mg on day 1 each 21-day cycle.
  Arms: Arm 2

SUMMARY:
Background:

Rare tumors of the genitourinary (GU) tract can appear in the kidney, bladder, ureters, and penis. Rare tumors are difficult to study because there are not enough people to conduct large trials for new treatments. Two drugs-sacituzumab govitecan (SG) and atezolizumab-are each approved to treat other cancers. Researchers want to find out if the two drugs used together can help people with GU.

Objective:

To test SG, either alone or combined with atezolizumab, in people with rare GU tumors.

Eligibility:

Adults aged 18 years and older with rare GU tumors. These may include high grade neuroendocrine carcinomas; squamous cell carcinoma of the bladder; primary adenocarcinoma of the bladder; renal medullary carcinoma; or squamous cell carcinoma of the penis.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have tests of heart function. They will have imaging scans. They may need a biopsy: A small needle will be used to remove a sample of tissue from the tumor.

Both SG and atezolizumab are given through a tube attached to a needle inserted into a vein in the arm.

All participants will receive SG on days 1 and 8 of each 21-day treatment cycle. Some participants will also receive atezolizumab on day 1 of each cycle.

Blood and urine tests, imaging scans, and other exams will be repeated during study visits.

Treatment may continue for up to 5 years.

Follow-up visits will continue for 5 more years.

DETAILED DESCRIPTION:
Background:

* Urothelial carcinoma (UC) represents the most common histology for tumors of the bladder and urinary tract.
* A minority of patients have primary tumors of the bladder/urinary tract consisting of rare histological variants, including high grade neuroendocrine carcinomas (HGNEC), primary adenocarcinoma of the bladder (urachal or non-urachal), or squamous cell carcinoma. Some tumors may contain elements of UC mixed with these variants or may be entirely composed of such variants.
* Clear cell renal cell carcinoma (ccRCC) is the most common histology for cancers of the renal parenchyma. Renal medullary carcinoma is a rare histology of kidney cancer, which is associated with sickle cell trait and other hemoglobinopathies.
* Rare tumors of the genitourinary (GU) tract often have more aggressive clinical course, but lack standard of care treatment regimens, since these patient populations are poorly represented or excluded from most clinical trials.
* Sacituzumab govitecan (SG) is an antibody-drug conjugate of an IgG 1 monoclonal antibody targeting trophoblastic cell surface antigen 2 (Trop2) with a chemotherapeutic payload of SN-38. SN-38 is an active metabolite of irinotecan and acts as a topoisomerase I inhibitor.
* SG has demonstrated clinical activity in solid tumors. In phase II clinical trials, SG has demonstrated efficacy in metastatic UC after progression on platinum-based chemotherapy and immune checkpoint inhibitor (ICI) therapy.
* Atezolizumab is an anti- programmed death-ligand 1 (PD-L1) ICI that is approved for advanced/metastatic UC in patients ineligible to receive platinum therapy.
* There are currently no clinical trials for SG monotherapy or SG/atezolizumab combination in rare GU tumors.

Objective:

-To determine clinical efficacy of sacituzumab govitecan (SG), either alone or in combination with atezolizumab, as defined by objective response rate (ORR), in participants with rare metastatic non-prostate genitourinary tumors

Eligibility:

* Age >= 18 years
* ECOG performance status <= 1
* Histologically confirmed diagnosis of locally advanced (unresectable) or metastatic GU tumors of the following histologies: high grade neuroendocrine carcinomas (HGNEC), squamous cell carcinoma, or primary adenocarcinoma of the bladder or urinary tract; or renal medullary carcinoma or squamous cell carcinoma of the penis.
* Participants must have locally advanced unresectable or metastatic disease on cross-sectional imaging.
* Participants may have received any prior programmed cell death protein 1 (PD-1)/PD-L1 axis ICI treatment.

Design:

* This is an open label, non-randomized phase II trial with two arms.
* All participants will receive SG.
* Participants without prior treatment with any PD-1/PD-L1 axis ICI (checkpoint inhibitor na(SqrRoot) ve) will be eligible to receive concurrent atezolizumab.
* SG will be administered intravenously (IV) at 10 mg/kg on D1 and D8 of 21-day cycles.
* Atezolizumab will be administered IV at 1200mg on D1 of 21-day cycles.
* Treatment will be given in 21-day cycles continuously for a maximum of 5 years, or until signs of progression or intolerable side effects.
* The accrual ceiling will be set at 60 to allow for inevaluable participants and screen failure.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically confirmed diagnosis of a locally advanced unresectable or metastatic non-prostate genitourinary (GU) tumor of the following histologies:

  * HGNEC, including, but not limited to, small cell carcinoma and large cell neuroendocrine carcinoma of the bladder or urinary tract
  * Squamous cell carcinoma of the bladder or urinary tract
  * Primary adenocarcinoma of the bladder or urinary tract (urachal or non-urachal)
  * Renal medullary carcinoma
  * Squamous cell carcinoma of the penis

Note: For the purposes of enrollment, the urinary tract is defined as the renal pelvis, ureter, bladder, and urethra.

* Pre-study treatment tissue availability (sufficient tissue for approximately 25 unstained slides is mandatory for enrollment. If tissue is determined to be insufficient/unsuitable, a fresh biopsy prior to study therapy will be required.
* Locally advanced unresectable or metastatic disease. Participants who have received prior treatment must have evidence of progressive disease (PD; i.e., defined as new or progressive lesions evident on cross-sectional imaging).
* Participants must have measurable disease, per RECIST 1.1.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky >= 70%.
* Adequate organ and marrow function as defined below:

  * Hemoglobin (Hgb) >= 9.0 g/dL
  * Absolute neutrophil count (ANC) >= 1,500/mcL
  * Platelets >= 100,000/mcL
  * Total bilirubin <= 1.5 x upper limit of normal (ULN) (<= 3 x ULN in participants with known/suspected Gilbert s disease)
  * AST/ ALT <= 2.5 x ULN (or <= 5 x ULN if considered to be related to liver metastases by the PI)
  * Serum creatinine <= 2 x ULN or creatinine clearance >= 30 ml/min/1.73 m^2 (glomerular filtration rate [GFR] may be used in place of CrCl. Creatinine clearance or eGFR should be calculated per institutional standard)
  * Alkaline phosphatase <= 2.5 x ULN (or <= 5 x ULN if considered to be related to liver or bone metastases by the PI)
  * Serum albumin >= 25g/L
  * For participants not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) <= 1.5 x ULN
  * For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* Participants may have received any number of prior anti-cancer treatments or be treatment na(SqrRoot) ve (except for participants with HGNEC of the bladder/urinary tract cancer, whom must have received a platinum-based combination regimen either as neoadjuvant, adjuvant or first-line treatment in the locally advanced/metastatic setting).
* Treated central nervous system (CNS) lesions, provided that all of the following criteria are met:

  * Measurable disease, per RECIST v1.1, must be present outside the CNS.
  * The participant has no history of intracranial hemorrhage or spinal cord hemorrhage.
  * The participant has not undergone stereotactic radiotherapy within 1 week prior to initiation of study treatment, whole-brain radiotherapy (WBXRT) within 2 weeks prior to initiation of study treatment, or neurosurgical resection within 4 weeks prior to initiation of study treatment.
  * The participant has no ongoing requirement for corticosteroids as therapy for CNS disease.
  * The participant may be receiving anti-convulsant therapy if appropriate and the dose is considered stable.

Prior treatment as follows:

* Prior radionuclide treatment must have a washout period of at least 6 weeks prior to the first dose of study treatment.
* Prior treatment with chemotherapy must have a washout period of 2 weeks prior to the first dose of study treatment.
* Prior treatment with non-CNS-directed radiotherapy must have a washout period of 2 weeks prior to the first dose of study treatment (except palliative bone-directed radiotherapy which does not require any washout).
* Prior treatment with a small molecule kinase inhibitor must have a washout period of at least 2 weeks or five half-lives of the compound or active metabolites, prior to the first dose of study treatment.
* Prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) must have a washout period of at least 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the first dose of study treatment.
* Major surgical procedure, other than for diagnosis, must not occur within 4 weeks prior to the first dose of study treatment.
* Prior treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) must have a washout period of at least 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Participants who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* FDA-approved hormonal therapy for the treatment or prevention of other malignancies (e.g., breast cancer, prostate cancer) are allowed to be continued where in the opinion of the treating investigator stopping such therapies may increase the risk of disease progression. Potential drug-drug interactions with the hormonal agent will be assessed by the treating investigator prior to enrollment and hormonal agents that inhibit or induce UGT1A1 will be excluded while on trial.
* Human immunodeficiency virus (HIV)-infected participants are eligible if on stable dose of highly active antiretroviral therapy (HAART), a CD4 count >= 200 cells/microL, and an undetectable viral load.
* Hepatitis B virus (HBV) positive participants are eligible if they have been treated or are on an appropriate course of antivirals at study entry and with planned monitoring and management according to appropriate guidance. For previously treated patients or those with prior infection that has been cleared, prophylaxis is permitted, and hepatology consultation recommended.
* Participants with a history of hepatitis C virus (HCV) infection (i.e., positive HCV antibody test) must have been treated and cured (negative HCV RNA test at screening). Participants with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
* Individuals of child-bearing potential (IOCBP) and individuals able to father a child must agree to use an effective method of contraception as follows:

  * IOCBP must agree to use one (1) highly effective methods of contraception (e.g., intrauterine device [IUD], hormonal, surgical sterilization) prior to study entry, for the duration of study participation, and for up to 6 months after discontinuation of the study drug(s). Participants must refrain from donating eggs during this same period.
  * Individuals able to father children must agree to use an effective method of contraception (barrier, surgical sterilization) for the duration of the study treatment and up to 6 months after the last dose of the study drug(s) and must refrain from donating sperm during this same period.
* Nursing participants must discontinue nursing and/or not begin nursing until 1 month after the last dose of study drug(s).
* Ability of participants to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of severe hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to SG, SN-38, irinotecan, or atezolizumab, or hypersensitivity to Chinese hamster ovary cell products.
* Symptomatic or untreated brain/CNS metastases.
* Positive serum or urine Beta-human chorionic gonadotropin (Beta-hCG) test at screening.
* Participants unwilling to accept blood products as medically indicated.
* Active or history of autoimmune disease or immune deficiency that might recur, which might affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These conditions include myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area.
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
    * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Anticipation of need for a major surgical procedure during the study.
* Prior allogeneic stem cell or solid organ transplantation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during SG or atezolizumab treatment or within 5 months after the final dose of SG or atezolizumab. Note: Seasonal flu vaccines that do not contain a live virus and locally authorized/approved COVID-19 vaccines are permitted.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) with the exception of participants with indwelling catheters (e.g., PleurX(R)) who are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN).
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, cerebrovascular accident, unstable arrhythmia, or unstable angina) within 3 months prior to initiation of study treatment.
* Prior treatment with immune checkpoint blockade therapies, including anti-PD-1, and anti-PD-L1 therapeutic antibodies (for Arm 2 only).
* Participants with prior malignancy within the previous 2 years except for locally curable cancers that have been apparently cured such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or low risk Gleason 6 prostate cancer, among others. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for the study.
* Participants with severe uncontrolled intercurrent illness that would limit compliance with study requirements, evaluated by history, physical exam, and chemistry panel.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | On days 1 and 8 of each cycle and at every restaging (every 9 weeks) until the end of the study therapy and every 9 weeks during follow-up until PD.
  Percentage of participants by best overall response (e.g., CR, PR, SD, PD) to therapy

SECONDARY OUTCOMES:
Duration of response (DoR) | On days 1 and 8 of each cycle and at every restaging (every 9 weeks) until the end of the study therapy and every 9 weeks during follow-up until PD.
  Time from start of treatment to disease progression or death in participants who achieve CR or PR
Overall survival (OS) | Days 1 and 8 of each cycle, at EoT, at the Safety visit, at follow-up, and every 90 days for up to a total of 5 years after the end of therapy
  Time from the start of treatment that participants are still alive.
Progression-free survival (PFS) | At every restaging (every 9 weeks) until the end of the study therapy and every 9 weeks during follow-up until PD
  Duration of time from start of treatment to time of progression or death, whichever occurs first
Clinical benefit rate (CBR) | At every restaging (every 9 weeks) until the end of the study therapy and every 9 weeks during follow-up until PD
  Percentage of participant who have achieved CR, PR, and SD while on treatment.
Safety of sacituzumab govitecan with or without atezolizumab | From first dose through 30 days after last treatment
  Adverse events (AEs) will be reported by type and grade of toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers at least 3 years after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- [Derived] Kydd AR, Chandran E, Simon NI, Atiq S, Ley L, Wang TF, Cordes L, Patel R, Smith E, Boudjadi S, Niglio SA, Yousefi-Rad A, Weng S, Stukes I, Banday AR, Akbulut D, Gurram S, Redd B, Steinberg S, Choo-Wosoba H, Apolo AB. A phase 2 study of sacituzumab govitecan with or without atezolizumab in rare genitourinary tumors (SMART) - design and rationale. Future Oncol. 2025 Aug;21(18):2261-2268. doi: 10.1080/14796694.2025.2516901. Epub 2025 Jun 23. PMID 40548513
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001535-C.html